CLINICAL TRIAL: NCT00297440
Title: Exercise to Aid Smoking Cessation in Adolescent Girls
Brief Title: Exercise, Smoking Cessation and Adolescents
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Temple University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Melissa Napolitano, PhD, Temple University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R03CA119712 (NIH)
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Smoking
Keywords: Smoking; Exercise; Adolescent; Girls
MeSH Terms: conditions — Smoking; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive-behavioral treatment
Behavioral: Exercise

SUMMARY:
We seek to: 1) conduct the formative work to adapt the cessation materials and exercise protocol from focus on adult women to adolescent girls, and 2) conduct a small randomized pilot trial to determine the preliminary efficacy of the intervention in a sample of adolescent girls. Therefore, this study, will serve as a pilot for a larger clinical trial. Successful smoking cessation in adolescent girls could contribute to the future reduction of chronic disease morbidity and mortality in this group.

DETAILED DESCRIPTION:
Approximately 22% of youth currently smoke cigarettes despite the increased risk of cancer and cardiovascular disease associated with cigarette use. Tobacco use continues to be the leading, preventable cause of mortality among US adults. Research has shown that those who smoke their first cigarette between the ages of 14-26 are more likely to become nicotine dependent, and, therefore, more resistant to smoking cessation efforts, than those initiating smoking at a later age. Although the smoking prevalence among girls declined in the 1970's and 1980's, the current smoking rates among high school girls has held constant from 1998 to 2000. Despite the negative health consequences associated with smoking, weight concerns and fear of weight gain have been shown to be associated with the uptake of smoking in girls. Alternatively, exercise has been shown to be a positive health behavior, and can provide the same perceived benefits of smoking: self-esteem, relaxation, weight management. In previous trials in adult women, vigorous intensity exercise has been shown to be effective for aiding with smoking cessation. Therefore, this study will adapt the efficacious group-based cognitive behavioral smoking cessation treatment plus exercise to meet the needs of adolescent girls. This project will consist of two phases. In Phase I of this project, 4 focus groups will be conducted (each consisting of 8-10 adolescent girls) to adapt the intervention. Adaptations will include making the materials, intervention content, and language age-appropriate and relevant for youth. Phase II of the project will consist of a randomized pilot study in which 40 adolescent girls will be randomly assigned to: a) standard cognitive-behavioral smoking cessation plus exercise (CBT+Exercise) or b) standard cessation with equal contact time (Standard+Contact). The sample will be recruited, treated for 12 weeks and followed for 3 months. Smoking cessation outcome (continuous abstinence) will be validated by saliva cotinine. Exercise adherence will be validated by attendance at supervised sessions, and objective monitoring. Secondary analysis of proposed theoretical mediators of behavior change will be conducted, including weight concerns and self-efficacy. The primary hypothesis is that girls in the CBT+Exercise group will have higher quit rates than girls in the Standard+Contact group. In summary, we seek to: 1) conduct the formative work to adapt the cessation materials and exercise protocol from a focus on adult women to adolescent girls, and 2) conduct a small randomized pilot trial to determine the preliminary efficacy of the intervention in a sample of adolescent girls. Therefore, this study will serve as a pilot for a larger clinical trial. Successful smoking cessation in adolescent girls could contribute to the future reduction of chronic disease mortality in this group.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent will be required for participation in the project

Exclusion Criteria:

* For Phase I of the study, we will recruit adolescent girls who report smoking at least 5 cigarettes per day for 6 months. We will recruit approximately 40 girls to participate in one of 4 focus groups. For Phase II, we will recruit adolescent female smokers (n = 40) aged 13-19. Potential participants for Phase II must smoke at least 5 cigarettes per day and be sedentary (i.e., participating in physical activity two days per week or less for 30 minutes or less each day). Other specific eligibility requirements for both phases include: a) having no physical or mental limitations that would restrict their ability to be active or complete study measures; b) passing the Physical Activity Readiness Questionnaire (PAR-Q).

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-08 (Actual); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Smoking status

SECONDARY OUTCOMES:
Physical Activity
Weight
Body image

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Napolitano, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States